CLINICAL TRIAL: NCT04341727
Title: Open-label, Randomized Controlled Trial of Hydroxychloroquine, Hydroxychloroquine Plus Azithromycin, Chloroquine Alone, Chloroquine Plus Azithromycin in the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS CoV-2) Infection
Brief Title: Hydroxychloroquine,Hydroxychloroquine,Azithromycin in the Treatment of SARS CoV-2 Infection
Acronym: WU352
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: DSMB recommended study suspension slow accrual
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jane O'Halloran, Assistant Professor in Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202003188
Record Dates: First submitted 2020-04-04; First posted 2020-04-10 (Actual); Results first posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections | interventions — Hydroxychloroquine; Azithromycin; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Hydroxychloroquine alone (Active Comparator): Arm 1: Hydroxychloroquine 400mg orally twice a day for one day, followed by 200mg twice a day for four consecutive days (Five days in total). The drug will be supplied in 200mg tablets.
  Interventions: Drug: Hydroxychloroquine Sulfate
- Hydroxychloroquine plus azithromycin (Active Comparator): Arm 2: Hydroxychloroquine 400mg orally twice a day for one day, followed by 200mg twice a day for four consecutive days (Five days in total). The drug will be supplied in 200mg tablets.
  AND Azithromycin 500mg orally once, followed by 250mg daily for four consecutive days (five days total). The drug will be supplied in 250mg tablets.
  Interventions: Drug: Hydroxychloroquine Sulfate; Drug: Azithromycin
- Chloroquine alone (Active Comparator): Arm 3: Chloroquine phosphate 1000mg orally once, followed in 12 hours by 500mg, then 500mg orally twice daily for 4 days (Five days in total). The drug will be supplied in 500mg tablets.
  Interventions: Drug: Chloroquine Sulfate
- Chloroquine plus azithromycin (Active Comparator): Arm 4: Chloroquine phosphate 1000mg orally once, followed in 12 hours by 500mg, then 500mg orally twice daily for 4 days (Five days in total). The drug will be supplied in 500mg tablets.
  AND Azithromycin 500mg orally once, followed by 250mg daily for 4 consecutive days (5 days total).The drug will be supplied in 250mg tablets.
  Interventions: Drug: Azithromycin; Drug: Chloroquine Sulfate

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate — anti-rheumatic drug (DMARD)
  Other Names: HYDROXYCHLOROQUINE Plaquenil
  Arms: Hydroxychloroquine alone; Hydroxychloroquine plus azithromycin
Drug: Azithromycin — Antibiotic
  Other Names: COMMON BRAND(S): Zithromax GENERIC NAME(S): Azithromycin
  Arms: Chloroquine plus azithromycin; Hydroxychloroquine plus azithromycin
Drug: Chloroquine Sulfate — Antimalarial
  Other Names: Aralen GENERIC NAME(S): Chloroquine Phosphate
  Arms: Chloroquine alone; Chloroquine plus azithromycin

SUMMARY:
This Phase III trial four treatment strategies non-critically ill hospitalized participants (not requiring intensive care unit (ICU) admission and/or mechanical ventilation) with SARS CoV-2 infection, Participants will receive hydroxychloroquine or chloroquine with or without azithromycin.

DETAILED DESCRIPTION:
This Phase III trial will utilize four treatment strategies in non-critically ill hospitalized participants (not requiring mechanical ventilation) with SARS CoV-2 infection, Participants will receive hydroxychloroquine or chloroquine with or without azithromycin. Investigators are primarily interested in the time to recovery. In addition to study medications there will be daily symptom surveys for 14 days, then weekly thereafter for 4 weeks resulting in a total duration of follow up of 42 days. During hospitalization, daily symptom surveys will be completed in conjunction with the study coordinators. On discharge participants will have the option to complete electronic symptom surveys or complete symptom surveys via telephone with study coordinator. In the event that the participant opts for electronic symptom surveys on discharge participants will in addition receive a follow up call from a study coordination every 7 days during the initial 14 day period. In addition, failure to submit a symptom survey will prompt a study follow up call. Data from standard of care SOC will be collected from medical records.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization for management of SARS CoV-2 infection
* Positive SARS CoV-2 test
* Age >=18 years
* Provision of informed consent
* Electrocardiogram (ECG) ≤48 hours prior to enrollment
* Complete blood count, glucose-6 phosphate-dehydrogenase (G6PD), comprehensive metabolic panel and magnesium ≤48 hours prior to enrollment from standard of care.
* If participating in sexual activity that could lead to pregnancy, individuals of reproductive potential who can become pregnant must agree to use contraception throughout the study. At least one of the following must be used throughout the study:

  * Condom (male or female) with or without spermicide
  * Diaphragm or cervical cap with spermicide
  * Intrauterine device (IUD)
  * Hormone-based contraceptive

Exclusion Criteria:

* Contraindication or allergy to chloroquine, hydroxychloroquine or azithromycin
* Current use hydroxychloroquine, chloroquine or azithromycin
* Concurrent use of another investigational agent
* Invasive mechanical ventilation
* Participants who have any severe and/or uncontrolled medical conditions such as:

  * unstable angina pectoris,
  * symptomatic congestive heart failure,
  * myocardial infarction,
  * cardiac arrhythmias or know prolonged QTc >470 males, >480 female on ECG
  * pulmonary insufficiency,
  * epilepsy (interaction with chloroquine),
* Prior retinal eye disease
* Concurrent malignancy requiring chemotherapy
* Known Chronic Kidney disease, eGFR<10 or dialysis
* G-6-PD deficiency, if unknown requires G6PD testing prior to enrollment

  * Known Porphyria
  * Known myasthenia gravis
  * Currently pregnant or planning on getting pregnant while on study
  * Breast feeding
  * AST/ALT >five times the upper limit of normal ULN*
  * Bilirubin >five times the ULN*
  * Magnesium <1.4 mEq/L*
  * Calcium <8.4mg/dL >10.6mg/dL*
  * Potassium <3.3 >5.5 mEg/L*

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-04-04 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane O'Halloran, MD PhD, Principal Investigator — Washington University School of Medicine (ID-CRU)
Locations (2):
- United States (2):
  - Washington University School of Medicine Infectious Disease Clinical Research Unit, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydroxychloroquine Plus Azithromycin: Arm 2: Hydroxychloroquine 400mg orally twice a day for one day, followed by 200mg twice a day for four consecutive days (Five days in total). The drug will be supplied in 200mg tablets.
  AND Azithromycin 500mg orally once, followed by 250mg daily for four consecutive days (five days total). The drug will be supplied in 250mg tablets.
  Hydroxychloroquine Sulfate: anti-rheumatic drug (DMARD)
  Azithromycin: Antibiotic
- Chloroquine Plus Azithromycin: Arm 4: Chloroquine phosphate 1000mg orally once, followed in 12 hours by 500mg, then 500mg orally twice daily for 4 days (Five days in total). The drug will be supplied in 500mg tablets.
  AND Azithromycin 500mg orally once, followed by 250mg daily for 4 consecutive days (5 days total).The drug will be supplied in 250mg tablets.
  Azithromycin: Antibiotic
  Chloroquine Sulfate: Antimalarial
Period: Overall Study
Arm/Group | Hydroxychloroquine Alone | Hydroxychloroquine Plus Azithromycin | Chloroquine Alone | Chloroquine Plus Azithromycin
Started | 9 | 7 | 7 | 7
Completed | 9 | 7 | 6 | 6
Not Completed | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxychloroquine Alone | Hydroxychloroquine Plus Azithromycin | Chloroquine Alone | Chloroquine Plus Azithromycin | Total
Number analyzed (Participants) | 9 | 7 | 7 | 7 | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [49 to 72] | 55 [48 to 60] | 54 [43 to 64] | 56 [44 to 62] | 55 [43 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 4 | 4 | 20
  Male | 2 | 2 | 3 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 8 | 4 | 7 | 6 | 25
  Unknown or Not Reported | 0 | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 5 | 4 | 18
  White | 4 | 2 | 2 | 3 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Hours to Recovery
Description: Time (hours) from randomization to recovery defined as 1) absence of fever, as defined as at least 48 hours since last temperature ≥ 38.0°C without the use of fever-reducing medications AND 2) absence of symptoms of greater than mild severity for 24 hours AND 3) not requiring supplemental oxygen beyond pre-COVID baseline AND 4) freedom from mechanical ventilation or death in each Arm/Group,respectively.
Time Frame: 42 days
Population: The sample size of 30 was well below the threshold for analysis
Measure: Mean (Inter-Quartile Range); unit: hours
Arm/Group | Hydroxychloroquine Alone | Hydroxychloroquine Plus Azithromycin | Chloroquine Alone | Chloroquine Plus Azithromycin
Number analyzed (Participants) | 9 | 7 | 7 | 7
hours | 96 [24 to 168] | 120 [48 to 240] | 168 [72 to 672] | 240 [48 to 288]

2. Secondary Outcome: Time to Fever Resolution
Description: Time to resolution of fever defined as at least 48 hours since last temperature ≥ 38.0°C without the use of fever-reducing medications in each Arm/Group,respectively.
Time Frame: 42 days
Population: The sample was well below the threshold for analysis
Measure: Mean (Inter-Quartile Range); unit: hours
Arm/Group | Hydroxychloroquine Alone | Hydroxychloroquine Plus Azithromycin | Chloroquine Alone | Chloroquine Plus Azithromycin
Number analyzed (Participants) | 9 | 7 | 7 | 7
hours | 72 [24 to 96] | 96 [48 to 120] | 72 [24 to 192] | 96 [48 to 144]

ADVERSE EVENTS:
Time Frame: 6 weeks per participant
Arm/Group | Hydroxychloroquine Alone | Hydroxychloroquine Plus Azithromycin | Chloroquine Alone | Chloroquine Plus Azithromycin
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 1/9 | 2/7 | 1/7 | 1/7
Other Adverse Events (participants affected / at risk) | 4/9 | 2/7 | 3/7 | 3/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine Alone (N=9) | Hydroxychloroquine Plus Azithromycin (N=7) | Chloroquine Alone (N=7) | Chloroquine Plus Azithromycin (N=7)
Pneumonia due to COVID (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Subject was previously discharged from hospital on room air . Subject came back to emergency department 4 days later with increased shortness of breath, secondary to COVID and readmitted
Urosepsis (Infections and infestations) | 0 (0) | 1 (4) | 0 (0) | 0 (0) — UTI the reason for the systemic shock
Respiratory Failure secondary to COVID (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Extended hospitalization due to worsening respiratory failure necessitating intubation and ECMO
Deep Vein Thrombosis- (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — hospitalization
Respiratory Failure secondary to Covid (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — requiring intubation
Bacterial Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Prolonged hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxychloroquine Alone (N=9) | Hydroxychloroquine Plus Azithromycin (N=7) | Chloroquine Alone (N=7) | Chloroquine Plus Azithromycin (N=7)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia due to COVID (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prolonged QtC (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blurred Vision (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory Failure due to Covid (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catatonia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatremia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prolonged QTc (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment in the clinical trial did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/27/NCT04341727/Prot_SAP_001.pdf